CLINICAL TRIAL: NCT01052142
Title: A Phase I Open-label Study of the Safety and Immunogenicity of Escalating Doses of Lipovaxin-MM, a Novel Melanoma Immunotherapeutic, in Patients With Metastatic Melanoma
Brief Title: Safety Study of a Liposomal Vaccine to Treat Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lipotek Pty Ltd (Industry)
Collaborators: Royal Adelaide Hospital (Other); Trident Clinical Research Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lipovaxin-MM-001
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Melanoma
Keywords: Melanoma; Cancer vaccines
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipovaxin-MM (Experimental)
  Interventions: Biological: Lipovaxin-MM

INTERVENTIONS:
Biological: Lipovaxin-MM — Patients will receive three doses of Lipovaxin-MM by intravenous infusion at intervals of four weeks OR patients will receive 4 doses of Lipovaxin-MM by intravenous infusion at weekly intervals

SUMMARY:
The purpose of this study is to determine whether Lipovaxin-MM, a new anti-cancer vaccine, is safe and effective in improving the body's ability to destroy cancer cells in patients with metastatic melanoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with incurable stage IV malignant melanoma for which no standard or curative therapy exist OR patients locoregionally recurrent melanoma (including local metastases, in transit metastases and satellitosis) where surgery is not the best therapeutic option.
* Must be able and willing to provide written informed consent.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Life expectancy of ≥12 weeks.
* Female subjects must be of non-child-bearing potential or using appropriate contraception.
* Positive test for cell mediated immunity.

Key Exclusion Criteria:

* Brain metastases or spinal cord compression, unless treatment was completed at least 4 weeks before entry and stable without steroid treatment for at least 4 weeks.
* Previous immunotherapy (except IL-2 or interferon-based therapy) for melanoma.
* Inadequate bone marrow reserve.
* Serum bilirubin ≥1.2 times the upper limit of normal.
* In absence of metastases, liver transaminase levels greater than 1.5 times the upper limit of normal.
* If metastases are evident, liver transaminase levels 2.5 times the upper limit of normal will be acceptable.
* Inadequate renal function.
* Evidence of severe or uncontrolled systemic diseases.
* Unresolved toxicity ≥CTC Grade 2 from previous anti-cancer therapy except alopecia (if applicable) unless agreed that the patient can be entered after discussion with the Medical Monitor.
* Participation in a trial of an investigational agent within the prior 30 days.
* HIV infection.
* Immunosuppressive therapy including corticosteroids within 4 weeks of screening.
* Pregnant or breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | Within 84 days after first dose
Immunogenicity | Within 42 days of first dose
  antigen specific immune responses will be monitored

SECONDARY OUTCOMES:
Anti-cancer activity (RECIST criteria) | Within 84 days of first dose
  assessed every 6 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brown, MBBS FRACP FRCPA, Principal Investigator — Royal Adelaide Hospital Cancer Centre
Locations (1):
- Pain & Anaesthesia Research Clinic, Adelaide, South Australia, Australia